CLINICAL TRIAL: NCT06291363
Title: Impact of Continuous Intraoperative Administration of Esmolol on Nociception Level-guided Control of Nociception. The EsmoNOL Randomized Controlled Trial
Brief Title: Impact of Administration of Esmolol on Nociception Level-guided Control of Nociception.
Acronym: ESMONOL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Pascal Laferrière-Langlois, MD, MSc, FRQS, Assistant Professor, Principal Investigator, Anesthesiologist, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-3612
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use, Unspecified; Anesthesia; Nociceptive Pain
Keywords: opioid sparing anesthesia; beta blockers; nociception monitoring; general anesthesia
MeSH Terms: conditions — Nociceptive Pain | interventions — esmolol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two groups of patients randomized into Group "ESMOLOL" for esmolol and group "Standard of Care" for a total of 64 participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done prior to the entrance in the OR, the day of the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esmolol (Experimental): In the Esmolol group, intravenous esmolol will be given as a bolus (0.5mg.kg-1) over 5 minutes, and will be started simultaneously to the remifentanil initiation.
  Once the bolus of esmolol is over, a perfusion of 20 mcg.kg-1.min-1 will be programmed and maintained until the end of the surgery and completion of skin sutures
  Interventions: Drug: Esmolol Hydrochloride
- Standard of care (Placebo Comparator): In the standard of care group, intravenous saline bolus, equivalent to an esmolol bolus (0.5mg.kg-1) will be given over 5 minutes, and will be started simultaneously to the remifentanil initiation.
  Once the bolus of saline is over, a saline perfusion equivalent to an esmolol infusion of 20 mcg.kg-1.min-1 will be programmed and maintained until the end of the surgery and completion of skin sutures
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Esmolol Hydrochloride — Patients in the experimental group will receive esmolol during general anesthesia
  Other Names: Brevibloc
  Arms: Esmolol
Drug: Saline — Patients in the standard of care group will receive saline as placebo during general anesthesia
  Other Names: saline serum
  Arms: Standard of care

SUMMARY:
This study aims to evaluate esmolol's perfusion impact during induction and maintenance of general anesthesia, using Nociception-Level-guided control of nociception, in adult patients undergoing laparoscopic and lower abdominal surgery, on intraoperative remifentanil consumption and postoperative pain in the Post-Anesthesia Care Unit.

DETAILED DESCRIPTION:
Opioids are currently the gold standard for perioperative pain control and allow for proper intraoperative hemodynamic stability. However, their use presents several major challenges, as demonstrated by the opioid crisis intensifying over the years in North America and increasingly in Europe. Besides commonly described adverse effects such as postoperative nausea, vomiting, respiratory depression, ileus, or pruritus, opioids are associated with induced hyperalgesia. In this context, several opioid-sparing strategies have been explored. The use of esmolol, a short-acting beta-blocker, can reduce sympathetic stimulation induced by perioperative nociceptive stimuli. Integrated into a multimodal strategy, it reduces the need for intraoperative opioid administration and postoperative analgesic consumption. Concurrently, multiparametric monitoring of nociception via the Nociception-Level Index (NOL index) also allows for a reduction in intraoperative opioids and decreased pain scores in the post anesthesia care unit (PACU).

The aim of this trial will be to explore the combination of these two strategies and assess the impact of continuous esmolol infusion on Nociception-Level-guided intraoperative remifentanil administration in patients under general anesthesia undergoing gynecological or general surgery via laparoscopy or lower abdominal laparotomy.

This single center randomized controlled trial will be conducted in a Canadian academic hospital. Participants aged between 18 and 65 years undergoing gynecological or general surgery by laparoscopy or lower abdominal laparotomy will be included in this study. Induction of general anesthesia will be achieved with propofol in combination with target-controlled infusion (TCI) remifentanil at 3 ng.ml-1 for intubation, then guided by the NOL Index during the procedure. Hypnosis will be maintained by the administration of sevoflurane with a target minimum alveolar concentration (MAC) between 0.7 and 1.2 to sustain a bispectral Index (BIS)between 40 and 60. Intervention group participants will receive esmolol as follows: an initial bolus of 0.5 mg.kg-1 at induction of anesthesia followed by a continuous infusion of 20mcg.kg-1.min-1 until the end of the intervention. A saline solution infusion will be administered to control group participants under the same conditions. The primary outcome will be the amount of remifentanil administered intraoperatively in mcg.kg-1.h-1. Secondary outcomes will include variations in the NOL Index during nociceptive stimuli, average heart rate and blood pressure, the intraoperative doses and time weighted average of norepinephrine (mg); ephedrine (mg), glycopyrrolate (mg) and atropine (mg), the total time and time weighted average of hypotension and or bradycardia during surgery, the time to first analgesic requirement, amount of morphine equivalent consumption for postoperative pain relief in PACU, intensity of pain at rest and under stress, using a verbal rating scale (VRS), from arrival to discharge from PACU.

The main objective of the study is to evaluate the impact of continuous intraoperative infusion of esmolol on intraoperative remifentanil administration in patients undergoing general anesthesia with NOL-guided nociception management.

Secondary objectives are listed below.

Based on a recent unpublished trial recently held at Maisonneuve-Rosemont Hospital focusing on colorectal surgeries, the investigators assumed a mean intraoperative remifentanil consumption of 5.59 mcg.kg-1.h-1 and 7.98, respectively in the intervention and control group, with a combined standard deviation of ± 3.24. This data is aligned with recently published international data. With an alpha risk of 5%, a power of 80.0%, a two-tailed test, and an estimated dropout ratio of 10.0%, it was calculated that 32 participants would be required in each group, to detect a 30% reduction in intraoperative remifentanil administration.

Study duration: 12 months

Study Center: Maisonneuve-Rosemont Hospital, Integrated University Health and Social Services Centre (CIUSSS) de l'Est de l'Ile de Montreal (CEMTL), University of Montreal, Montreal, Quebec, Canada.

Adverse Events: there is very little risk involved with participation in this study, side effects that may be associated with the use of esmolol includes bradycardia and/or hypotension

ELIGIBILITY:
Inclusion Criteria:

* Fully consented, American Society of Anesthesiologists Classification Score 1-3 patients from 18yo to 65yo
* Undergoing laparoscopic surgery associated with sub umbilical mini-laparotomy. Eligible surgeries will be hysterectomy (excluding vaginal approach) and left hemicolectomy, of duration time expected under 180 minutes, under general anesthesia
* No allergy to one of the medications used in this study

Exclusion Criteria:

Contraindication to the use of the study drug (esmolol) is an exclusion criterion :

* Hypotension
* Sinus bradycardia
* Sick sinus syndrome
* Second and third degree A-V block
* Pulmonary hypertension
* Right ventricular failure secondary to pulmonary hypertension
* Decompensated heart failure
* Cardiogenic shock
* Nontreated pheochromocytoma
* Known hypersensitivity to esmolol or any of the inactive ingredients of the product
* Allergy to esmolol or other beta blockers (cross-sensitivity is possible)
* Renal dysfunction
* Airway disease such as asthma or chronic obstructive pulmonary disease
* Thyrotoxicosis
* Myasthenia gravis
* Raynaud's disease or peripheral circulatory disorder

Other situations leading to exclusion :

* Severe mental impairment
* Chronic use of opioids, β-adrenergic receptors antagonists
* High risk of conversion to laparotomy according to the surgical team (>25%)

Patients will automatically be excluded after recruitment if they withdraw their consent, or if laparoscopy is converted to laparotomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-03-03 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
Intra operative remifentanil administration | intraoperative (from T0 = incision until Tend = end of dressing)
  Quantity of remifentanil in mcg.kg-1.h-1, administered between the first surgical incision and its discontinuation at wound dressing

SECONDARY OUTCOMES:
The NOL Index variation before and after orotracheal intubation and first surgical incision | intraoperative (from T0 = nociceptive stimulation Tend = 3 minutes post stimulation)
  The NOL Index variation before and after orotracheal intubation and first surgical incision
The mean intraoperative blood pressure and heart rate | intraoperative (from T0 = incision until Tend = end of dressing)
  The mean intraoperative blood pressure and heart rate during surgery
doses and time weighted of norepinephrine (mg); ephedrine (mg), glycopyrrolate (mg) and atropine (mg) | intraoperative (from T0 = incision until Tend = end of dressing)
  doses and time weighted average of norepinephrine (mg); ephedrine (mg), glycopyrrolate (mg) and atropine (mg)
Total time with NOL value above > 25 | intraoperative (from T0 = incision until Tend = end of dressing)
  Total time and time weighted average with NOL value above > 25
The total time and time weighted average of hypotension and/or bradycardia | intraoperative (from T0 = incision until Tend = end of dressing)
  The total time and time weighted average of hypotension (< 20% of the baseline values of the pre-anesthesia mean arterial pressure (MAP) and/or bradycardia (HR < 60 beats/min, or HR < 50 beats/min for a profound bradycardia)) during surgery
The time to first analgesic requirement in PACU | postoperative (from T0 = PACU arrival until Tend = PACU discharge)
  The time to first analgesic requirement in PACU
The amount of morphine equivalent consumption | postoperative (from T0 = PACU arrival until Tend = PACU discharge)
  The amount of morphine equivalent consumption for postoperative pain relief in the post anesthesia care unit (PACU) in both groups
The intensity of pain at rest and under stress | postoperative (from T0 = PACU arrival until Tend = PACU discharge)
  The intensity of pain at rest and under stress, using a verbal rating scale from 0 to 10 : 0 being no pain, and 10 the worst pain imaginable. I'll be assessed every 30 minutes from arrival to discharge from PACU
Postoperative nausea and vomiting (PONV) and antiemetics use | postoperative (from T0 = PACU arrival until Tend = PACU discharge)
  Postoperative outcomes such as postoperative nausea and vomiting (PONV) and amount of antiemetics used in PACU
The time spent in PACU | postoperative (from T0 = PACU arrival until Tend = PACU discharge)
  time spent in PACU (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Laferrière-Langlois, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Île de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Background] Asouhidou I, Trikoupi A. Esmolol reduces anesthetic requirements thereby facilitating early extubation; a prospective controlled study in patients undergoing intracranial surgery. BMC Anesthesiol. 2015 Nov 28;15:172. doi: 10.1186/s12871-015-0154-1. PMID 26615516
- [Background] Bergeron C, Brulotte V, Pelen F, Clairoux A, Belanger ME, Issa R, Urbanowicz R, Tanoubi I, Drolet P, Fortier LP, Verdonck O, Fortier A, Espitalier F, Richebe P. Impact of chronic treatment by beta1-adrenergic antagonists on Nociceptive-Level (NOL) index variation after a standardized noxious stimulus under general anesthesia: a cohort study. J Clin Monit Comput. 2022 Feb;36(1):109-120. doi: 10.1007/s10877-020-00626-4. Epub 2021 Jan 4. PMID 33398545
- [Background] Bohringer C, Astorga C, Liu H. The Benefits of Opioid Free Anesthesia and the Precautions Necessary When Employing It. Transl Perioper Pain Med. 2020;7(1):152-157. PMID 31712783
- [Background] Celebi N, Cizmeci EA, Canbay O. [Intraoperative esmolol infusion reduces postoperative analgesic consumption and anaesthetic use during septorhinoplasty: a randomized trial]. Rev Bras Anestesiol. 2014 Sep-Oct;64(5):343-9. doi: 10.1016/j.bjan.2013.10.013. Epub 2014 Jun 21. Portuguese. PMID 25168439
- [Background] Colvin LA, Bull F, Hales TG. Perioperative opioid analgesia-when is enough too much? A review of opioid-induced tolerance and hyperalgesia. Lancet. 2019 Apr 13;393(10180):1558-1568. doi: 10.1016/S0140-6736(19)30430-1. PMID 30983591
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Gelineau AM, King MR, Ladha KS, Burns SM, Houle T, Anderson TA. Intraoperative Esmolol as an Adjunct for Perioperative Opioid and Postoperative Pain Reduction: A Systematic Review, Meta-analysis, and Meta-regression. Anesth Analg. 2018 Mar;126(3):1035-1049. doi: 10.1213/ANE.0000000000002469. PMID 29028742
- [Background] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185
- [Background] Paloheimo MP, Sahanne S, Uutela KH. Autonomic nervous system state: the effect of general anaesthesia and bilateral tonsillectomy after unilateral infiltration of lidocaine. Br J Anaesth. 2010 May;104(5):587-95. doi: 10.1093/bja/aeq065. Epub 2010 Mar 30. PMID 20354006
- [Background] Renaud-Roy E, Stockle PA, Maximos S, Brulotte V, Sideris L, Dube P, Drolet P, Tanoubi I, Issa R, Verdonck O, Fortier LP, Richebe P. Correlation between incremental remifentanil doses and the Nociception Level (NOL) index response after intraoperative noxious stimuli. Can J Anaesth. 2019 Sep;66(9):1049-1061. doi: 10.1007/s12630-019-01372-1. Epub 2019 Apr 17. PMID 30997633
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Sabourdin N, Burey J, Tuffet S, Thomin A, Rousseau A, Al-Hawari M, Taconet C, Louvet N, Constant I. Analgesia Nociception Index-Guided Remifentanil versus Standard Care during Propofol Anesthesia: A Randomized Controlled Trial. J Clin Med. 2022 Jan 11;11(2):333. doi: 10.3390/jcm11020333. PMID 35054027
- [Background] Shahiri TS, Richebe P, Richard-Lalonde M, Gelinas C. Description of the validity of the Analgesia Nociception Index (ANI) and Nociception Level Index (NOL) for nociception assessment in anesthetized patients undergoing surgery: a systematized review. J Clin Monit Comput. 2022 Jun;36(3):623-635. doi: 10.1007/s10877-021-00772-3. Epub 2021 Nov 16. PMID 34783941
- [Background] Shanthanna H, Ladha KS, Kehlet H, Joshi GP. Perioperative Opioid Administration. Anesthesiology. 2021 Apr 1;134(4):645-659. doi: 10.1097/ALN.0000000000003572. PMID 32991672

DOCUMENTS (1):
  • Study Protocol (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT06291363/Prot_000.pdf